CLINICAL TRIAL: NCT01449734
Title: Observational Study of Family Satisfaction in the Intensive Care Unit Using the German-language FS-ICU
Brief Title: Family Satisfaction (FS) in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Center for Sepsis Control and Care, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Christiane Hartog, Principal investigator, Center for Sepsis Control and Care, Germany
Other Study IDs: Jena FS-ICU
Record Dates: First submitted 2011-09-30; First posted 2011-10-10 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-09

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is increasing awareness that high-quality care in the intensive care unit also includes care of visiting family members according to their needs. The investigators therefore want to assess family satisfaction using a questionnaire that was specially developed for this setting and recently validated for German-speaking participants.

DETAILED DESCRIPTION:
Family members who visit patients on the ICU (intensive care unit) are not just onlookers. They experience the process of care along with their loved ones. Increasingly, the satisfaction of family members with ICU care, decision-making and information, and their empowerment to contribute towards patient care as near relatives, is being perceived as an important aspect of the general quality of ICU care.

Family satisfaction is assessed using the 34-item FS-ICU questionnaire which was recently validated for German-speaking participants.

The aim of this pilot survey is to identify opportunities for improvement of family satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* all visiting family members who consent to participate

Exclusion Criteria:

* no more than two family members per patient;
* prior participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Visiting family members of patients being treated in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane S Hartog, MD, Principal Investigator — Jena University Hospital, Dpt. of Anesthesiology and Intensive Care Medicine
Locations (1):
- Intensive Care Units of the University Hospital Jena, Jena, Thuringia, Germany

REFERENCES:
- [Background] Wall RJ, Engelberg RA, Downey L, Heyland DK, Curtis JR. Refinement, scoring, and validation of the Family Satisfaction in the Intensive Care Unit (FS-ICU) survey. Crit Care Med. 2007 Jan;35(1):271-9. doi: 10.1097/01.CCM.0000251122.15053.50. PMID 17133189
- [Background] Heyland DK, Rocker GM, Dodek PM, Kutsogiannis DJ, Konopad E, Cook DJ, Peters S, Tranmer JE, O'Callaghan CJ. Family satisfaction with care in the intensive care unit: results of a multiple center study. Crit Care Med. 2002 Jul;30(7):1413-8. doi: 10.1097/00003246-200207000-00002. PMID 12130954
- [Background] Stricker KH, Kimberger O, Schmidlin K, Zwahlen M, Mohr U, Rothen HU. Family satisfaction in the intensive care unit: what makes the difference? Intensive Care Med. 2009 Dec;35(12):2051-9. doi: 10.1007/s00134-009-1611-4. PMID 19730813
- [Derived] Schwarzkopf D, Behrend S, Skupin H, Westermann I, Riedemann NC, Pfeifer R, Gunther A, Witte OW, Reinhart K, Hartog CS. Family satisfaction in the intensive care unit: a quantitative and qualitative analysis. Intensive Care Med. 2013 Jun;39(6):1071-9. doi: 10.1007/s00134-013-2862-7. Epub 2013 Feb 16. PMID 23417207
- See also: Publication of study results — http://www.ncbi.nlm.nih.gov/pubmed/23417207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective cohort study performed in four (mixed surgical, neurological, and cardiological) intensive care units of a university hospital in Germany
Groups:
- Family Satisfaction: family satisfaction in the intensive care unit (ICU) and areas for improvement
Period: Overall Study
Arm/Group | Family Satisfaction
Started | 215
Completed | 215
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Visiting family members
Arm/Group | Family Satisfaction
Number analyzed (Participants) | 215
Age, Customized [Number; unit: participants] — Numbers in categories do not add to 215 because of non-response.
  participants
    18-34 | 11
    35-44 | 28
    45-54 | 55
    55-64 | 55
    > 64 | 60
Gender [Number; unit: participants] — Gender of participating relatives. Numbers do not add to 215 because of non-response.
  participants
    Female | 136
    Male | 62

OUTCOME MEASURES:

1. Secondary Outcome: Patient Severity of Illness
Time Frame: From beginning of ICU stay until death or discharge of patient, whatever came first, assessed up to 2 months
Reporting Status: Not Posted

2. Secondary Outcome: Patient Length of Stay on the ICU
Time Frame: From beginning of ICU stay until death or discharge of patient, whatever came first, assessed up to 2 months
Reporting Status: Not Posted

3. Secondary Outcome: Patient Mortality
Time Frame: From beginning of ICU stay until death or discharge of patient, whatever came first, assessed up to 2 months
Reporting Status: Not Posted

4. Primary Outcome: Family Satisfaction in the ICU (FS-ICU) Questionnaire- Overall Satisfaction Score
Description: Overall satisfaction score is calculated as the mean of 24 Items concerning satisfaction with care, communication and decision-making. After transformation of Items the score has a scale reaching from 0 (highly unsatisfied) to 100 (highly satisfied).
Time Frame: From beginning of ICU stay until death or discharge of patient, whatever came first, assessed up to 2 months
Population: By invitation
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family Satisfaction: All 215 surveyed relatives are contained in this group, since the study was observational without intervention.
Arm/Group | Family Satisfaction
Number analyzed (Participants) | 215
units on a scale | 78.3 (14.3)

ADVERSE EVENTS:
Time Frame: March to November 2011
Description: No adverse events were expected by conducting the survey among family members of ICU patients. Thus adverse events were not assessed.
Arm/Group | Family Satisfaction
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes